CLINICAL TRIAL: NCT03423225
Title: A Single Center, Single Arm, Open-label Study to Evaluate the Efficacy and Safety of Tacrolimus Modified Release, ADVAGRAF® After Treatment With a Tacrolimus in New Liver Transplant Recipients
Brief Title: To Evaluate the Efficacy and Safety of ADVAGRAF® After Treatment With a Tacrolimus in New Liver Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kim, Seoung-Hoon (Other Government)
Collaborators: Astellas Pharma Korea, Inc. (Industry); Linical Korea (Industry)
Responsible Party: Sponsor-Investigator, Kim, Seoung-Hoon, Head of Organ transplantation department, National Cancer Center, Korea
Organization: National Cancer Center, Korea (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Assign
Record Dates: First submitted 2018-01-22; First posted 2018-02-06 (Actual); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Liver Transplantation
Keywords: ADVAGRAF®; Liver Transplantation; tacrolimus
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ADVAGRAF® (Experimental): One arm: Treatment conversion will take placefrom twice daily tacrolimus to once daily tacrolimus (ADVAGRAF) 3 months after transplant in new liver transplant recipients.
  Interventions: Drug: ADVAGRAF®

INTERVENTIONS:
Drug: ADVAGRAF® — Administration method The total daily dose of tacrolimus will be converted to 1:1 (mg:mg) and the total daily dose of ADVAGRAF® will be administered only once daily in the morning, starting from Day 1 (at least one hour before breakfast or 2 to 3 hours after breakfast).
  * Dose adjustment after conversion On Day 1, the total dose will be converted to 1:1. It is recommended to check the blood concentration of tacrolimus at each visit and adjust the dose to achieve the blood concentration maintaining at 5~8ng/ml for 0 to 3 months and then at 5ng/ml or below for 3 to 6 months of study treatment.
  * Duration of treatment The investigational product will be administered for 24 weeks.
  Other Names: tacrolimus

SUMMARY:
This study's objective is to evaluate the incidence rate of acute rejection reactions after 24 weeks treatment with ADVAGRAF® following 3 months treatment with tacrolimus in new liver transplant recipients.

Treatment conversion will take place from twice daily tacrolimus to once daily tacrolimus (ADVAGRAF) 3 months after transplant in new liver transplant recipients.

DETAILED DESCRIPTION:
This is single center,open-label study with ADVAGRAF® Primary endpoint is Incidence rate of biopsy confirmed acute rejection reactions within 24 weeks following conversion+ Incidence rate of acute rejection reactions (%) = number of subjects with at least one acute rejection reaction 1)/total number of subjects in the relevant analysis set * 100 Only those acute rejection reactions confirmed by biopsy will be acceptable as acute rejection reactions.

Administration method is following The total daily dose of tacrolimus will be converted to 1:1 (mg:mg) and the total daily dose of ADVAGRAF® will be administered only once daily in the morning, starting from Day 1 (at least one hour before breakfast or 2 to 3 hours after breakfast).

* Dose adjustment after conversion On Day 1, the total dose will be converted to 1:1. It is recommended to check the blood concentration of tacrolimus at each visit and adjust the dose to achieve the blood concentration maintaining at 5~8ng/ml for 0 to 3 months and then at 5ng/ ml or below for 3 to 6 months of study treatment.
* Duration of treatment The investigational product will be administered for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. When the Subjects agree informed consent form, Subject should be More than 20 years of age
2. Those who was transplanated liver at a minimum of 10 weeks or Maximum of 14 weeks before the baseline
3. Average of tacrorimus minimum blood concenration level is 3-10 ng/mL from transplanted date to baseline.
4. Female subjects who have child bearing potential must have a negative at urine or serum pregnancy test prior to enrollment and must agree to practice effective contraceptive measures during the study.(The oral contraceptive pill is not allowed to take a female subject)
5. Subjects who are clinically stable judged by investigator.
6. Subjects capable of understanding the purpose and risks of the study, having been fully informed and has given written informed consent to participate in the study

Exclusion Criteria:

1. Subjects previously received an organ transplantation excluding liver transplantation. Or Subjects received an auxiliary graft or bioartificial liver(cell system).
2. Recently there was acute rejection from the day of liver transplantation to baseline
3. If the onset of a new malignant cancer after liver transplantation is diagnosed, well treated basal cell carcinoma or squamous cell carcinoma is classified as an exception
4. When it is known that there is a hypersensitivity reaction to the ingredients of tacrolimus or the test drug
5. In the opinion of the investigator, there is an unstable medical condition that can affect the purpose of the clinical trial
6. In the event of material abuse, mental disorder or anything that can not smoothly communicate with the inverstigator in the opinion of the investigator
7. Currently, if subjects are participating in other clinical trials or if subjects receive another drug for clinical trials within 28 days before baseline
8. If subjects have received a prohibited combination therapy currently or within 28 days before the baseline
9. Pregnant or lactating women
10. If known for HIV-positive
11. When there is a high possibility that subject will not be able to obey the visit schedule planned in protocol
12. Those who have clinically significant renal dysfunction judged by the investigator or at baseline serum creatinine level exceeds 1.6 mg / dL or GFR (MDRD) is less than 30 mL / min
13. Those who have clinically significant liver function disorder judged by the investigator or at the baseline, the values of SGPT / ALT and / or SGOT / AST and / or bilirubin are more than three times the upper limit of the laboratory normal range When raised

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-03-22 (Actual); Primary Completion 2017-07-18 (Actual); Study Completion 2017-12-14 (Actual)

PRIMARY OUTCOMES:
Incidence rate of acute rejection reaction confirmed by biopsy within 24 weeks after conversion | within 24 weeks
  Incidence rate of acute rejection reaction (%) = The number of subjects with at least one acute rejection reaction / Total number of subjects included in the analysis group * 100 number of subjects in the relevant analysis set * 100

SECONDARY OUTCOMES:
Severity of acute rejection reaction confirmed by biopsy within 24 weeks after conversion | within 24 weeks
  Severity of acute rejection reactions is defined as the highest severity in a subject who had at least one acute rejection reaction.
Survival rates of subjects after conversion | at week 24
Survival rate of transplanted organs after conversion | at week 24
Blood concentration of tacrolimus | at week -4, week 0, week 2, week 4, week 8, week 16 and week 24

CONTACTS AND LOCATIONS:
Overall Officials: Seoung-Hoon Kim, doctoral, Principal Investigator — National Cancer Center, Republic of Korea

IPD SHARING:
Plan to Share IPD: No